CLINICAL TRIAL: NCT03385499
Title: TOXODIAG: New Diagnostic Approach for Congenital Toxoplasmosis
Brief Title: New Diagnostic Approach for Congenital Toxoplasmosis
Acronym: TOXODIAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A02208-45
Record Dates: First submitted 2017-11-03; First posted 2017-12-28 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Congenital Toxoplasmosis
Keywords: Congenital toxoplasmosis; Neonatal biological diagnosis of congenital toxoplasmosis; neonatal diagnosis; ELISPOT; IgG
MeSH Terms: conditions — Toxoplasmosis, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- negative control group (Other): blood additional samples on negative control group
  Interventions: Biological: blood additional samples
- positive control group (Other): blood additional samples on positive control group
  Interventions: Biological: blood additional samples
- seroconversion group (Other): blood additional samples on seroconversion group
  Interventions: Biological: blood additional samples

INTERVENTIONS:
Biological: blood additional samples — additional samples of mother's blood and umbilical cord at delivery

SUMMARY:
Caused by Toxoplasma gondii, toxoplasmosis is mostly asymptomatic except in immunocompromised individuals and infants infected in utero. Congenital toxoplasmosis (CT) results from the transplacental passage of the parasite, which occurs in 30% of cases of primary infection during pregnancy. Neonatal biological diagnosis of toxoplasmosis is essential in the case of (i) suggestive clinical signs in the newborn with no information on the serological status of the mother, (ii) seroconversion diagnosed during pregnancy, (iii) not or poorly followed pregnancy, and (iiii) for enhanced effectiveness of treatments administered as soon as possible to the newborn. Given the limitations of current diagnostic tests, the characterization of specific immunoglobulin (Ig)G neo-synthesized by the newborn would be of great help for an early diagnosis of CT.

The main objective of the TOXODIAG project is to validate and evaluate the ELISPOT (Enzyme-Linked Immunosorbent SPOT assay) method for detecting, in the newborn, B lymphocytes (LyB) sensitized in utero to produce T. gondii specific immunoglobulins (Ig) following a primary infection of the mother during the pregnancy. More precisely, the detection and quantification of LyB secreting IgG and IgM specific for T. gondii using the ELISPOT method will be applied i) to mononuclear cells of women in seroconversion following a toxoplasmic primo-infection during pregnancy and ii) to cord blood mononuclear cells of newborns suspected of CT, in comparison to positive and negative infection controls.

To reach this goal, TOXODIAG is a diagnostic, multicentric, prospective, non-randomized, comparative and controlled study. It will be performed in 3 parallel groups of pregnant women performing prenatal follow-up and giving birth in the maternity wards of 3 hospitals of the AP-HP (Louis MOURIER, Bichat-Claude Bernard and Cochin) which ensure mother/child follow-up and biological sampling, with great gynecology and obstetrics expertise. Sixty women will be selected and included into 3 groups according to toxoplasmic seroconversion during pregnancy (n=30), positive (n=15) or negative (n=15) toxoplasma serology. The necessary biological material will consist in additional blood tubes which will be taken at the same time as those performed for the usual pregnancy follow-up examinations and will correspond to maternal peripheral blood at inclusion, seroconversion and delivery as well as cord blood.

DETAILED DESCRIPTION:
Toxoplasmosis is a cosmopolitan parasitosis that affects one third of the world's population. This infection, caused by Toxoplasma gondii, is mostly asymptomatic except in immunocompromised individuals and infants infected in utero. Congenital toxoplasmosis (CT) results from the transplacental passage of the parasite, which occurs in 30% of cases of primary infection during pregnancy. The clinical consequences are all the more serious when fetal contamination is early (death in utero, premature delivery or term childbirth with perivisceral involvement) and result in mainly neuro-ocular attacks in case of later contamination. Pregnant women or women of childbearing age therefore constitute a group at risk and are exposed differently according to their geographical situation and food consumption. Neonatal biological diagnosis of toxoplasmosis is essential in the case of (i) suggestive clinical signs in the newborn with no information on the serological status of the mother, (ii) seroconversion diagnosed during pregnancy, (iii) not or poorly followed pregnancy, and (iiii) for enhanced effectiveness of treatments administered as soon as possible to the newborn. This diagnosis is based mainly on parasite research in the neonatal amniotic fluid or placenta by PCR and / or inoculation in mice, as well as on serological tests. Immunoglobulins (Ig) A and IgM do not cross the placental barrier and represent good markers of congenital infection in the newborn. Nevertheless, they are not specific to an acute infection and are no longer detectable at birth in cases of infections contracted by the mother before the 3rd trimester of pregnancy. The detection of IgG synthesized by the child has a diagnostic value only after 6 months of life, once the materno-transmitted IgG have been eliminated, and the techniques comparing the IgG response profiles of the mother and the child to a plurality of toxoplasmic antigens remain difficult to interpret (western blot, ELIFA). It is nevertheless a combination of these different tests that makes up the decision tree for a neonatal biological diagnosis of CT. The characterization of specific IgG neo-synthesized by the newborn would be of great help for an early diagnosis of congenital infection by T. gondii. The present project consists in determining the presence in the neonate of B lymphocytes (LyB) sensitized in utero to produce specific IgG in case of CT. This approach can be envisaged because of the maturity acquired by the fetal LyB from the end of the first trimester of pregnancy, demonstrated by their ability to produce high affinity Ig in the case of maternal infection or neonatal immunization.

This research is diagnostic, multicentric, prospective, non-randomized, comparative and controlled. It will be performed in 3 parallel groups of pregnant women performing prenatal follow-up and giving birth in the maternity wards of 3 hospitals of the AP-HP which ensure mother/child follow-up and biological sampling, with great gynecology and obstetrics expertise. Sixty patients will be selected and included according to the following distribution:

* Positive control group (women with positive toxoplasma serology): 15 patients;
* Negative control group (women with negative toxoplasma serology): 15 patients;
* Group of women diagnosed with toxoplasmic seroconversion during pregnancy: 30 patients.

Non-recruiting centers will be HUPC and HUPNVS biology laboratories for the realization of serological tests and expertise in biological diagnosis and IRD UMR 216 for coordination, laboratory experiments and expertise in immunology.

ELIGIBILITY:
Inclusion Criteria:

In all cases, pregnant women whose age ≥ 18 years are concerned.

* Seroconversion group: a diagnosis of toxoplasmic seroconversion will be documented by a negative serology in early pregnancy which becomes positive during pregnancy, with the synthesis of specific IgG;
* Positive control group: known and documented positive toxoplasmosis serology;
* Negative control group: known and documented negative serology for toxoplasmosis at 7 months of pregnancy.

Exclusion Criteria:

Non-inclusion criteria common to the three groups

* Expected delivery in another maternity that does not participate in the study;
* Positive serology for HIV;
* Contra-indication to additional tubes during the blood sampling corresponding to the usual follow-up of pregnancy (anemia, all other case according to the evaluation of the clinician in charge of the follow-up);
* Absence of social insurance or CMU or AME;
* Vulnerable pregnant woman (under guardianship or curatorship);
* No signature of consent to participate in research.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 60 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Detection/quantification of T. gondii IgG and IgM secreting LyB by ELISPOT on cord blood mononuclear cells (MNC) of newborns suspected of congenital toxoplasmosis. | 6 months
  Umbilical cord blood will be collected at birth. A circuit is put in place to ensure a transfer to the research lab in order to assess the MNC isolation under 24 hours after blood drawing. Isolated MNC are thereafter frozen at -80°C until realization of the ELISPOT assay, using the adaptation of the test as validated under the Secondary Outcome Measures 1, 4 and 5 (test duration; multiple Ig detection; impact of the type of T. gondii capture antigen).

SECONDARY OUTCOMES:
Detection/quantification of T. gondii IgG and IgM secreting LyB by ELISPOT on mononuclear cells (MNC) of pregnant women with toxoplasma primary infection. | 6 months
  Peripheral blood will be collected in the maternities of the study. Isolated MNC will be frozen at -80°C until realization of the ELISPOT assay, with a focus on two main adjustments: lowering form 7 to 2 the number of days of duration of the test; simultaneous detection of IgM and IgG.
Comparison of the number of T. gondii IgG and IgM secreting LyB revealed by ELISPOT between the three groups of mothers at delivery: positive control group, negative control group and seroconversion group. | 6 months
  Peripheral blood will be collected in the maternities of the study. Isolated MNC will be frozen at -80°C until realization of the ELISPOT assay, with expected results according to the T. gondii serological status at delivery.
Comparison of the number of T. gondii IgG and IgM secreting LyB revealed by ELISPOT in mothers at time of the seroconversion biological diagnosis and at delivery. | 6 months
  Peripheral blood will be collected in the maternities of the study. Isolated MNC will be frozen at -80°C until realization of the ELISPOT assay, with an evaluation of the kinetics of anti-T. gondii IgM and IgG secreting cells.
Comparison of the number of specific IgG and IgM secreting LyB revealed by ELISPOT in T. gondii primary infected-mothers at their delivery and in their newborns. | 6 months
  Maternal peripheral blood as well as cord blood will be collected in the maternities of the study. Isolated MNC will be frozen at -80°C until realization of the ELISPOT assay, with an evaluation of the maturity of the infant's immune system. This will be done by comparing the patterns of the LyB cell spots of a mother and her infant, with indication on both affinity and avidity.
Comparison of the number of T. gondii IgG and IgM secreting LyB revealed by ELISPOT performed using either T. gondii type I or type II as capture antigen. | 6 months
  Demonstration of ubiquity of the ELISPOT assay applied to T. gondii IgM and IgG detection: ubiquity will be demonstrated if numbers of secreting B cells are not different.
Comparison of the diversity of LyB cell populations between groups of women (toxoplasma infected or not during pregnancy) and infants (suspected of toxoplasma congenital infection or not). | 6 months
  Molecular study using the Ig spectratyping technique, in order to investigate the Ig variable region specialized in antigen recognition : it will allow to highlight the LyB populations which have been sensitized by T. gondii.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Migot Nabias, PhD, Principal Investigator — university Paris Descarte
Locations (3):
- France (3):
  - Hopital Louis Mourier, Colombes
  - Hopital Bichat, Paris
  - Hopital Cochin, Paris

IPD SHARING:
Plan to Share IPD: Undecided